CLINICAL TRIAL: NCT04579289
Title: Managerial and Environmental Risk for COVID 19 in French Long Term Care Institutions_COVID-19
Brief Title: Managerial and Environmental Risk for COVID 19 in French Long Term Care Institutions
Acronym: REMPAR-EHPAD
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8898_REMPAR-EHPAD
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: Covid19; Elderly; Long term care; Crisis Management; France
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — A questionnaire was e-mailed to all identified institutions, with 3 reminders in one month. It included 39 questions concerning :
  * morbidity and mortality linked with COVID-19
  * structural features of the facility (location, architecture, residents characteristics)
  * human resources
  * crisis management (visits and circulation restrictions, personal protective equipment)

SUMMARY:
REMPAR EHPAD study addresses environmental and managerial factors associated with an outbreak of COVID 19 in French Long Term Care Institutions in the spring of 2020. The survey used a mixed methodology, combining qualitative and quantitative approaches, with a questionnaire send to all identified institutions (n=501) and qualitative interviews with facility directors (n=21).

DETAILED DESCRIPTION:
1. Declarative retrospective survey :

   A questionnaire was e-mailed to all identified institutions, with 3 reminders in one month. It included 39 questions concerning :
   * morbidity and mortality linked with COVID-19
   * structural features of the facility (location, architecture, residents characteristics)
   * human resources
   * crisis management (visits and circulation restrictions, personal protective equipment) A statistical analysis by logistic regression will be made, to identify explanatory variables for the occurrence of at least one COVID 19 infection among the residents.
2. Qualitative survey :

The investigators conducted semi-directed face-to-face interviews with facility directors. The investigators realized a purposive sample to assure maximal variability of the facilities (location, size, status, severity of the outbreak). The interview guide focused on structural, organizational, and human factors at stake in outbreak management, to identify incentives and obstacles associated with an easier crisis management.

ELIGIBILITY:
Inclusion Criteria:

* Long Term Care Institution (EHPAD) in Britain, France,

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Long Term Care Institution (EHPAD) director
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
case of COVID 19 | 01 september 2020, survey closing date
  Number of case (confirmed or probable) of COVID 19 in each facility

CONTACTS AND LOCATIONS:
Overall Officials: Aline MD CORVOL, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France